CLINICAL TRIAL: NCT04493138
Title: Phase I/II Study of Azacitidine in Combination With Quizartinib for Patients With Myelodysplastic Syndromes and Myelodysplastic/Myeloproliferative Neoplasms With FLT3 or CBL Mutations
Brief Title: Azacitidine and Quizartinib for the Treatment of Myelodysplastic Syndrome or Myelodysplastic/Myeloproliferative Neoplasm With FLT3 or CBL Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1178; NCI-2020-05261 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1178 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Recurrent Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Azacitidine; quizartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (azacitidine, quizartinib) (Experimental): Patients receive azacitidine SC or IV over about 30 minutes on days 1-5 and quizartinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Quizartinib

INTERVENTIONS:
Drug: Azacitidine — Given SC or IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Quizartinib — Given PO
  Other Names: AC-220; AC010220; AC220

SUMMARY:
This phase I/II trial studies the side effects and best dose of quizartinib when given with azacitidine and to see how well they work in treating patients with myelodysplastic syndrome or myelodysplastic/myeloproliferative neoplasm with FLT3 or CBL mutations. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Quizartinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving azacitidine and quizartinib may help to control myelodysplastic syndrome or myelodysplastic/myeloproliferative neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and maximum tolerable dose (MTD) of quizartinib in combination with azacytidine.

II. To assess overall response (ORR) rate to quizartinib in combination with azacitidine.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS), duration of response, leukemia-free survival (LFS), relapse-free survival (RFS) and safety profile.

II. Correlative studies.

OUTLINE: This is a phase I, dose-escalation study of quizartinib followed by a phase II study.

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over about 30 minutes on days 1-5 and quizartinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years as MDS is a very rare disease in the pediatric setting.
2. Diagnosis of MDS or MDS/MPN including CMML according to WHO.
3. For hypomethylating agent naïve patients: int-2 or higher by IPSS or >5% bone marrow blasts if MDS or dysplastic CMML (WBC <13x109/L). Patients with proliferative (WBC >/= 13x109/L) CMML or MDS/MPN, or those with dysplastic CMML with high-risk molecular features (mutations in ASXL1, TP53 or more than 3 mutations) are also eligible independently of IPSS risk score or bone marrow blast percentage.
4. For patients with prior hypomethylating agent therapy: no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 or relapse or progression after any number of cycles.
5. Detectable FLT3-ITD mutation in bone marrow and/or peripheral blood, or presence of CBL exon 8 or 9 deletions or point mutations.
6. Serum creatinine </= 2xULN.
7. Adequate hepatic function with total bilirubin <2x ULN (will allow less than 5xULN if Gilbert's at investigator's discretion), AST or ALT </=3xULN.
8. ECOG Performance Status 0-2.
9. Patient must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study.
10. Prior hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (eg, G-CSF, GM-CSF, procrit, aranesp, thrombopoietins) is allowed at any time prior to or during study if considered to be in the best interest of the patient.

Exclusion Criteria:

1. Uncontrolled infection not adequately responding to appropriate antibiotics.
2. Screening ECG with a QTcF >450 msec. The QTcF interval will be calculated by Fridericia's correction factor (QTcF). The QTcF will be derived from the average QTcF in triplicate. Patients are excluded if they have QTcF >450. Subjects with prolonged QTcF interval in the setting of RBBB (right bundle branch block) may participate upon review and approval by the principal investigator and following evaluation by cardiology consult.
3. Patients with congenital long QT syndrome.
4. History or presence of sustained ventricular tachycardia requiring medical intervention.
5. Any history of clinically significant ventricular fibrillation or torsades de pointes.
6. Known history of second- or third-degree heart block (may be eligible if the patient currently has a pacemaker).
7. Sustained heart rate of <50/minute on screening ECG. The heart rate will be derived from the average heart rate in triplicate.
8. Right bundle branch block + left anterior hemiblock (bifascicular block).
9. Complete left bundle branch block.
10. Atrial fibrillation documented within 2 weeks prior to first dose of study drug.
11. New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <50 by echocardiogram or multigated acquisition (MUGA) scan.
12. History of myocardial infarction within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias.
13. Patients who are actively taking a strong CYP3A4 inducing medication
14. Patients who require treatment with concomitant drugs that prolong QT/QTc interval or strong CYP3A4 inhibitors with the exception of antibiotics, antifungals, and antivirals that are used as standard of care to prevent or treat infections, antiemetics (such as ondansetron) and other such drugs that are considered absolutely essential for the care of the subject or if the Investigator believes that beginning therapy with a potentially QTc-prolonging medication (such as anti-emetic) is vital to an individual subject's care while on study.
15. Female patients who are pregnant or lactating.
16. Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermidical jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study.
17. Female patients with reproductive potential who do not have a negative urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening.
18. Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy.
19. Patients known to be positive for hepatitis B surface antigen expression or with active hepatitis C infection (positive by polymerase chain reaction or on antiviral therapy for hepatitis C within the last 6 months). Patients with history of HIV disease are also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At least 4 cycles of therapy in the absence of progression (1 cycle = 28 days)
  Will be defined as complete remission, partial remission, complete remission with incomplete count recovery, marrow compete remission or hematological improvement. Will be estimated for all patients along with the 95% credible interval.
Overall survival | Time from treatment start till death or last follow-up, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator.
Duration of response | Duration from the first documented onset of partial response or complete response to the date of progressive disease/relapse, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator.
Relapse-free survival | Time from start of response to the date of event defined as the first documented progressive disease/relapse or death, whichever comes first, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator.
Leukemia free survival | Time from treatment start to the time of progression to leukemia or death, assessed up to 2 years
  Will be listed and summarized by the Kaplan-Meier estimator.
Incidence of adverse events (AEs) | Up to 2 years
  The severity of the toxicities will be graded according to the latest version of National Cancer Institute Common Terminology Criteria for Adverse Events. The number and percent of subjects with treatment-emergent adverse events will be summarized according to intensity and drug relationship, and categorized by System Organ Class and preferred term by dose level/Part. All reported AEs that occur after signing informed consent will be included in the analysis of all reported AEs. Exposure to study drug and reasons for discontinuation of study drug will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Bravo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Montalban-Bravo G, Jabbour E, Chien K, Hammond D, Short N, Ravandi F, Konopleva M, Borthakur G, Daver N, Kanagal-Shammana R, Loghavi S, Qiao W, Huang X, Schneider H, Meyer M, Kantarjian H, Garcia-Manero G. Phase 1 study of azacitidine in combination with quizartinib in patients with FLT3 or CBL mutated MDS and MDS/MPN. Leuk Res. 2024 Jul;142:107518. doi: 10.1016/j.leukres.2024.107518. Epub 2024 May 11. PMID 38744144
- See also: http://www.mdanderson.org — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT04493138/ICF_000.pdf